CLINICAL TRIAL: NCT04229706
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Study on the Efficacy and Safety of Xiangjurupining Capsule in the Treatment of Hyperplasia of Breast (Liver Stagnation and Phlegm Coagulation)
Brief Title: A Study of Xiangjurupining Capsule in the Treatment of Hyperplasia of Breast (Liver Stagnation and Phlegm Coagulation)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-XJRPNJN-Ⅱ
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Hyperplasia of Breast
Keywords: hyperplasia of breast; Xiangjurupining capsule
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose group (Experimental): xiangjurupining capsule ,8 capsules，tid
  Interventions: Drug: High dose Xiang Ju Ru Pi Ning capsule
- Lower dose group (Experimental): xiangjurupining capsule, 4 capsules,tid, xiangjurupining capsule placebo ,4 capsules，tid，po
  Interventions: Drug: Low dose Xiang Ju Ru Pi Ning capsule
- Placebo group (Placebo Comparator): xiangjurupining capsule placebo ,8 capsules，tid，po
  Interventions: Drug: Xiang Ju Ru Pi Ning capsule placebo

INTERVENTIONS:
Drug: High dose Xiang Ju Ru Pi Ning capsule — xingjurupining capsule,8 capsule,tid,3 months.
  Other Names: High dose group
  Arms: High dose group
Drug: Low dose Xiang Ju Ru Pi Ning capsule — xiangjurupining capsule,4 capsules , and xiangjurupining capsule placebo,4 capsules,tid,3 months.
  Other Names: Low dose group
  Arms: Lower dose group
Drug: Xiang Ju Ru Pi Ning capsule placebo — xiangjurupining capsule,8 capsule,tid,3 months.
  Other Names: Placebo group
  Arms: Placebo group

SUMMARY:
The study is to evaluate the efficacy and safety of two doses of xiangjurupining capsule in Hyperplastic disease of breast patients .

DETAILED DESCRIPTION:
The study is to evaluate the efficacy and safety of two doses of xiangjurupining capsule,give three times a day versus placebo in Hyperplastic disease of breast patients .The clinical phase of the study comprises a run-in period，an 3-months double-blind treatment period and a 1-month follow-up period, resulting in 5-months overall duration of the study for each patient.

Patients report their breast pain as measured using NRS scale on the subject daily diary。

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-50 years.
2. Those who meet the diagnostic criteria of breast hyperplasia and has a course of more than 3 months;
3. Conform to the syndrome differentiation standard of liver depression and phlegm coagulation;
4. Patients have a basic regular menstrual cycle (21-35 days) and a menstrual period (3-7 days)
5. BI-RADS grade 2-3
6. NRS score ≥ 4 points in screening period
7. The average score of NRS was ≥ 4 in the run-in period, and there was still a target lump in palpation
8. Volunteer to participate in the experiment and sign the informed consent form after informed consent（Patients voluntarily accepted the test and gave informed consent）

Exclusion Criteria:

1. Patients with other breast diseases or other causes of breast pain, such as mastitis, breast cancer, etc.
2. Patients with severe cardiovascular and cerebrovascular diseases, liver, kidney, malignant tumor, blood system diseases and mental diseases.
3. Patients who have been confirmed with dysfunctional uterine bleeding, amenorrhea, polycystic ovary syndrome, menopausal syndrome and hyperprolactinemia before, still need to be treated by regulating hormone level.
4. Patients with previously confirmed hypercortisolism who still need to be treated with bromocriptine.
5. Those with menstrual period more than 7 days, menopause and serious irregular menstrual cycle.
6. Alt, AST, ALP, TBIL, GGT more than 1.2 times the upper limit of normal value; serum Cr, bun more than 1.2 times the upper limit of normal value, or blood, urine routine, ECG and other examination items are abnormal and of clinical significance.
7. That who pregnant or lactating women, or have a pregnant plan within the next 6 months
8. Chinese or Western medicine was used to treat hyperplasia of mammary gland within 1 month before the treatment and during run-in period(including external application medicine, acupuncture, etc.) and hormone drugs have been used within half a year (except for long-term oral contraceptives).
9. Allergic constitution, known to be allergic to the ingredients of the prescription of the test drug
10. History of alcohol or drug abuse.
11. Participants in other clinical trials within 3 months before screening
12. According to the judgment of the researchers, there are other diseases or situations that reduce the possibility of enrollment or complicate the enrollment, such as frequent changes in the working environment, which are likely to cause lost visits, and people with mental and behavioral disorders that cannot be based on the full informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
The pain of breast | up to 3 months
  Subject reported breast pain using NRS( Numerical Rating Scale)scale on the subject daily diary..The NRS scale is a line composed of 11 points, marked with a scale of 0 to 10. The subjects rated themselves according to the most painful degree every day. The higher the score, the higher the degree of pain.
The days of pain | up to 3 months
  Subject reported breast pain as measured using NRS scale on the subject daily diary.The number of the pain days was calculated and compared with the baseline which the number of pain days in the lead-in period.
The target lump | 3 months after treatment
  Assess the scope ,the size and the hardness of the target lump by palpation.The doctor palpated the breast of the subjects and measured the size of the target lump with a ruler.Four quadrant method was used to record the number of the target lump's quadrants.Four level（0,2,4,6） to measure The scope,the size and the hardness of lump .the Score from 0(none) to 6(most severe).
The target lump area | 3 months after treatment
  Assess the breast glandular section thickness, breast duct width and nodules of the target lump area by B-ultrasound.
TCM syndrome scores | 3 months after treatment
  Compared wth baseline,the scores of changes of TCM syndrome Evaluation at each visit .This instrument consists of two primary symptoms: breast pain, breast mass ,and four secondary symptoms.Four levels to measure severity of primary symptoms（0、2、4、6）and secondary symptoms（0、1、2、3）, respectively. Record the tongue and pulse conditions. The TCM syndrome effect calculated by nimodipine method. The final score has a range of 0 to 100. The effect of TCM syndrome from 0% (negative ) to 100% (disappear).

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Baoding No.1 Hospital of TCM, Baoding
  - Dongfang Hospital ,Beijing University of Chinese Medicine, Beijing
  - Dongzhimen Hospital,Beijing University of Chinese Medicine, Beijing
  - Guangdong Provincial Hospital of TCM, Guangzhou
  - the First Affiliated Hospital of Guangzhou University of TCM, Guangzhou
  - Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai
  - SHUGUANG Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai
  - Weifang Traditional Chinese Hospital, Weifang